CLINICAL TRIAL: NCT02896244
Title: AssessmeNT of the Incidence of Clostridium Difficile Infections in Hospitalized Patients on Antibiotic TrEatment
Acronym: ANTICIPATE
Status: Completed | Type: Observational
Sponsor: MJM Bonten (Other)
Collaborators: Da Volterra (Industry); Universitätsklinikum Köln (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor-Investigator, MJM Bonten, Professor of molecular epidemiology of infectious diseases, head of department of medical microbiology, UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: COMBACTE WP7
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Clostridium Difficile
Keywords: Clostridium difficile; Clostridium difficile infection; antibiotics; antibiotics associated diarrhea; microbiome; microbiota
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial DNA from rectal swab samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention

SUMMARY:
During or after antibiotic treatment, antibiotic residues impair the intestinal microbiota (gut flora) and lead to adverse effects such as the emergence of bacterial resistance or the occurrence antibiotic-associated diarrhoea (AAD) including antibiotic-induced C. difficile infection (CDI). The spread of resistant Gram-negative bacteria and the increasing number and severity of CDI are considered as worldwide public health threats.

Da Volterra is a biotechnology company developing a novel product, DAV132 (a medical device in Europe), intended to prevent these antibiotic adverse effects. Da Volterra is planning to carry out a phase 2-3 randomized controlled trial (RCT) of DAV132 in the prevention of antibiotic-induced CDI. The RCT will involve hospitalized patients aged ≥50 years old and treated with predefined antibiotic classes known to increase the risk of CDI. The incidence of CDI in this population is unknown, yet, incidence is an important determinant for the required sample size.

Therefore, the main objective of the current study is to assess CDI incidence in patients ≥50 years of age treated with predefined antibiotic classes.

In addition, to optimise the target population of the DAV132 RCT, the effect of the predefined antibiotic agents on the intestinal microbiota will be assessed. Furthermore, biomarkers predictive of CDI occurrence might help identify patients at high risk for the disease, which could further optimise the RCT. No validated biomarkers have been described in the literature yet. Assessment of potential biomarkers is another aim of the present study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female hospitalized patient.
2. Aged ≥ 50 years old.
3. Initiation of intravenous or oral treatment with intended duration ≥5 days (≥1 day for clindamycin) with at least one of the following antibiotic classes, or treatment scheduled within the next 72 hours:

   * Third or fourth generation cephalosporins
   * Fluoroquinolones
   * Penicillins +beta-lactamase inhibitors
   * Clindamycin
   * Carbapenems
4. Written informed consent provided prior to inclusion.

Exclusion Criteria:

1. Ongoing antibiotic treatment with one of the above classes initiated >6 hours before inclusion into the study.
2. ICU admission at the time of inclusion or anticipated admission within 48h.
3. Suspected or diagnosed CDI, ongoing treatment for CDI, or diarrhoea at the time of inclusion.
4. Patient with stoma.
5. Subject has been included into this study previously.
6. Patient treated with probiotics to prevent CDI.
7. Patient with any social or logistical condition which in the opinion of the investigator may interfere with the conduct of the study, such as incapacity to well understand, not willing to collaborate, or cannot easily be contacted after discharge.
8. Subject is subject to legal protection.
9. Subject deprived of liberty by judicial or administrative decision.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 50 or older receiving oral or intervenous antibiotic treatment with Third or fourth generation cephalosporins, Fluoroquinolones, Penicillins +beta-lactamase inhibitors, Clindamycin, or Carbapenems during hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Clostridium difficile infection | 28 days

SECONDARY OUTCOMES:
Clostridium difficile infection | 90 days
Antibiotics associated diarrhea | 90 days
Bacterial diversity | 6 days
  Change from baseline to day 6 of bacterial diversity and composition of the intestinal microbiome
Urine sulfate levels | 6 days
  Change from baseline to day 6 of 3-indoxyl sulfate levels in urine (corrected for the urine creatinine levels)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bonten, MD, PhD, Principal Investigator — UMC Utrecht
Locations (34):
- France (8):
  - CHD Vendee, La Roche-sur-Yon
  - CHU Dupuytren, Limoges
  - APHP Beaujon, Paris
  - APHP Bichat, Paris
  - APHP Hôpital Cochin, Paris
  - Hôpital St Louis, Paris
  - CH de Cornouaille, Quimper
  - Centre Hospitalier Universitaire de Tours, Tours
- Germany (8):
  - Uniklinik der RWTH, Aachen
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Essen, Essen
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - UK Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Lübeck
  - Klinikum der Universität München, München
- Greece (5):
  - Evangelismos General Hospital of Athens, Athens
  - Ippokratio Hospital of Athens, Athens
  - Laiko General Hospital, Athens
  - University General Hospital ATTIKON, Athens
  - University Hospital of Heraklion, Irakleio
- University Medical Center, Utrecht, Netherlands
- Romania (5):
  - Infectious and Tropical Diseases Hospital "Dr. Victor Babes", Bucharest
  - The National Institute of Infectious Diseases Matei Bals, Bucharest
  - Cluj Napoca Infectious disease Clinical Hospital, Cluj-Napoca
  - Oncology Institute Ion Chiricuta Cluj Napoca, Cluj-Napoca
  - Clinical Hospital Of Infectious Diseases Of Iasi, Iași
- Spain (7):
  - Bellvitge Hospital, Barcelona
  - Hospital Universitari Vall d´Hebrón, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No
16S rRNA and shotgun metagenomic sequence data generated and analyzed in this study have been deposited in the NCBI Sequence Read Archive with the accession code PRJNA685914. Human reads were identified and removed prior to shotgun metagenomics data upload. Access to clinical data is restricted as the informed consent provided does not allow for use of clinical data outside the research institution. Data are available from the corresponding author upon reasonable requests.

REFERENCES:
- [Result] van Werkhoven CH, Ducher A, Berkell M, Mysara M, Lammens C, Torre-Cisneros J, Rodriguez-Bano J, Herghea D, Cornely OA, Biehl LM, Bernard L, Dominguez-Luzon MA, Maraki S, Barraud O, Nica M, Jazmati N, Sablier-Gallis F, de Gunzburg J, Mentre F, Malhotra-Kumar S, Bonten MJM, Vehreschild MJGT; ANTICIPATE Study Group. Incidence and predictive biomarkers of Clostridioides difficile infection in hospitalized patients receiving broad-spectrum antibiotics. Nat Commun. 2021 Apr 14;12(1):2240. doi: 10.1038/s41467-021-22269-y. PMID 33854064
- [Result] Berkell M, Mysara M, Xavier BB, van Werkhoven CH, Monsieurs P, Lammens C, Ducher A, Vehreschild MJGT, Goossens H, de Gunzburg J, Bonten MJM, Malhotra-Kumar S; ANTICIPATE study group. Microbiota-based markers predictive of development of Clostridioides difficile infection. Nat Commun. 2021 Apr 14;12(1):2241. doi: 10.1038/s41467-021-22302-0. PMID 33854066
- See also: COMBACTE consortium website: ANTICIPATE is WP7 of COMBACTE — https://www.combacte.com/trials/anticipate/